CLINICAL TRIAL: NCT05023538
Title: PROTECTION Study: PReventiOn of HearT Failure in Type 2 Diabetes by ExerCise InTerventION
Brief Title: Prevention of Heart Failure in Type 2 Diabetes by Exercise Intervention
Acronym: PROTECTION
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hasselt University (Other)
Collaborators: Jessa Hospital (Other); KU Leuven (Other); University Ghent (Other)
Responsible Party: Principal Investigator, Dominique Hansen, Professor, Hasselt University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Version 1, 10/06/2021
Record Dates: First submitted 2021-06-24; First posted 2021-08-26 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Type 2 Diabetes
Keywords: T2D; exercise; rehabilitation; training; global longitudinal strain; echocardiography; heart; cardiac remodelling
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Motor Activity

STUDY DESIGN:
Intervention Model Description: Single-blind randomized controlled trial and a cohort study.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Researchers performing the outcome assessments and analyses will be blinded to treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Usual care (No Intervention): No intervention
- Low-volume moderately-intense exercise (Experimental): exercise at 50-65%VO2peak; 20-30min/training session, 3x/week, 6 months
  Interventions: Other: Cycling
- High-volume moderately-intense exercise (Experimental): exercise at 50-65%VO2peak; 20-50min/training session, 3x/week, 6 months
  Interventions: Other: Cycling
- Low-volume high-intense exercise (Experimental): exercise at 50-85%VO2peak; 20-30min/training session, 3x/week, 6 months
  Interventions: Other: Cycling

INTERVENTIONS:
Other: Cycling — Exercise on bicycle ergometer
  Arms: High-volume moderately-intense exercise; Low-volume high-intense exercise; Low-volume moderately-intense exercise

SUMMARY:
Global longitudinal strain emerged as an important predictive marker that could be assessed during echocardiography. It enabled the detection of subclinical myocardial systolic dysfunction, without observable reductions in cardiac output or left ventricular ejection fraction, often years before diabetes induced heart failure. In asymptomatic T2D patients with no history of cardiovascular disease, an impaired global longitudinal strain is a predictor of future adverse left ventricular remodeling and adverse cardiovascular events. Exercise training is a promising intervention to interfere in the diabetes induced heart failure pathophysiology. However, the impact of different exercise modalities (e.g. intensity and volume) on the global longitudinal strain in type 2 diabetes (T2D) is unknown.

DETAILED DESCRIPTION:
More than 400 million people worldwide are affected by diabetes mellitus whose prevalence keeps increasing. In type 2 diabetes mellitus (T2DM), up to 23% of the patients have asymptomatic diastolic and 13% systolic cardiac dysfunction. Diabetes-induced heart failure (DIHF), with reduced or preserved ejection fraction, is thus one of the major complications of T2DM, which is characterized by structural and functional changes in the myocardium in absence of coronary artery disease, other cardiac pathologies or hypertension. These changes significantly affect prognosis: patients with DIHF are at a 147% elevated risk for premature death within 4 years vs. 29% in patients without DIHF. It is thus of the utmost importance to prevent the development of DIHF. Although the exact mechanisms are not fully understood, hyperglycemia, hyperinsulinemia and hyperlipidemia are considered as key risk factors, but also oxidative and dicarbonyl stress, advanced glycation end products (AGEs) and inflammation play an important role in the pathophysiology of DIHF.

To prevent adverse cardiac remodeling in T2DM and the development of DIHF, early biomarkers are mandatory. In this respect, in the past few years global longitudinal strain (GLS) emerged as an important predictive marker that could be assessed during echocardiography: the global longitudinal strain enables the detection of subclinical myocardial systolic dysfunction, without observable reductions in cardiac output or left ventricular ejection fraction, often years before DIHF. In asymptomatic T2DM patients with no history of cardiovascular disease, an impaired GLS is a predictor of future adverse left ventricular (LV) remodeling and adverse cardiovascular events, thus providing incremental prognostic value beyond clinical data, glycated hemoglobin (HbA1c) and diastolic function. The investigators found that GLS is indeed significantly lowered (by ±14%, at rest and during low-intense and high-intense exercise, in asymptomatic well-controlled T2DM patients (HbA1c: 6.9±0.7%). During exercise, GLS increases in T2DM, but fails to normalize when compared with healthy controls. In contrast to current assumption, the investigators' data demonstrate that a disturbed GLS is highly common in T2DM patients.

Exercise training is strongly recommended to T2DM patients, and is a crucial treatment next to medication and diet, as this (further) optimizes glycemic control by improving insulin sensitivity, next to the positive impact on physical fitness, blood pressure, lipid profile and body composition. Recent evidence also indicates a significantly lowered mortality in habitual physically active vs. non-active T2DM patients (hazard ratio=0.61).

What type of exercise is most effective? What remains debatable is whether exercise intervention can prevent the development of DIHF in asymptomatic T2DM patients. According to a recent systematic review from the investigators' laboratory, the impact of exercise intervention on GLS in asymptomatic T2DM is equivocal: significant improvements from some studies could not be reproduced in other. In line with these findings, the investigators' unpublished pilot data also reveal the capability of exercise training to improve GLS in some T2DM patients.

The investigators' data show the potency of exercise in preventing DIHF in asymptomatic T2DM patients, but they also show that crucial aspects deserve further study to maximize the benefits of exercise training on GLS in T2DM patients, and hereby to offer maximal protection against the development of DIHF.

The impact of different exercise modalities (e.g. intensity, volume) on GLS in T2DM patients is currently unknown. In the only clinical study that examined T2MD patients to date, results show that high-intense interval training is more effective to improve GLS, as opposed to moderate-intense exercise training. However, the study is biased due to the lack of supervision in the moderate-intense trained group and the lack of control for equal caloric expenditure between training groups. Therefore, it is likely that differences in exercise volume could be at the basis of different changes in GLS between groups. Indeed, the investigators' pilot data, in which iso-caloric interventions were compared, show different results: moderate-intense exercise training seems more potent to improve GLS, as opposed to high-intense interval training. As a result, although there is evidence that exercise training improves GLS in T2DM patients, it remains to be studied whether different volumes or intensities are of key importance.

Despite following identical exercise interventions, studies and the investigators' pilot data also show significant inter-subject variances in changes in GLS. Therefore, the impact of the patient's phenotype, as well as habitual physical activity (PA) and dietary habits, on the effects of exercise training on GLS in T2DM patients is currently unknown. Revealing which (non-)modifiable patient-related factors (e.g. phenotype, habitual PA and dietary habits) predict the responsiveness of GLS to exercise intervention in T2DM patients may lead to a more patient-specific application of such intervention or further tailoring of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* physically inactive (no participation in structured or unstructured physical activity (PA) and not reaching the recommended PA guidelines: initially based on the International Physical Activity Questionnaire )
* age between 30-75 years
* blood HbA1c of 6-10% (if taking blood glucose lowering medication) or 6.5-10% without taking blood glucose lowering medication, and/or two-hour plasma glucose ≥11.1 mmol/L or ≥200 mg/dL following a 75g oral glucose load during OGTT.
* women of child bearing age will be included into the trial.

Exclusion Criteria:

* exogenous insulin therapy
* individuals suffering from any disease with significant impact on exercise intervention participation, such as: chronic heart disease or significant arrhythmias, cardiac events (myocardial infarction, coronary artery bypass graft, percutaneous coronary intervention), chronic obstructive pulmonary, cerebrovascular or peripheral vascular disease, severe hypertension (>160/110 mmHg), cancer, severe neuropathy (limiting exercise participation).

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — 1:1 men/women distribution
Enrollment: 182 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
mPAP/CO and mPAP/CO slope | at baseline and 6 months
  * Mean pulmonary artery pressure by cardiac output and by cardiac output slope
  * mPAP/CO slope will be calculated via measurement of LVOTdiameter, LVOT VTI and sPAP at three timepoints during exercise echocardiography. These timepoints are: rest, low intense exercise (HR<100 before fusion of early and late mitral inflow (E & A)), and high-intense exercise (RER 1.02-1.05).
Global longitudinal strain (%) | at baseline and 6 months
  Cardiac function evaluation by echocardiography at rest

SECONDARY OUTCOMES:
Fasted Blood draw | baseline, 3m and 6m
  lipid profile (HDL, LDL, triglicerides, free fatty acids, total cholesterol) glycemic profile (Hba1c, fasting glucose and insulin) kidney function (eGFR, creatinine)
Cardiopulmonary exercise testing on a bicycle | baseline, 3m and 6m
  Peak CPET values:
  Load, HR, VE, Bf, SBP, DBP, VO2, VCO2, RER, VE/VCO2, VE/VO2, SpO2, PETCO2, PETO2, BR
Rest and exercise echocardiography | baseline and 6m
  Supine resting echocardiography
  * Structure (LVOTd, IVSd, LVEDD, PWd, RWT, LVMI)
  * Function (LVOT VTI, LVEDV biplane, LVESV biplane, Evel, A vel, e' sep, e' lat, VCI exp, VCI ins, RAP, TR velocity, TRPG, PASP, GLS, TAPSE, LAVI)
  Semisupine exercise echocardiography at rest, low-intensity exercise (HR<100) and high-intensity exercise (RER 1.2-1.05)
  - Function (LVOT VTI, RVAd, RVAs, TAPSE, MAPSE, LVEDV biplane, LVESV biplane, LVEF, Evel, Avel, e'sep, e'lat, LV s'sep, LV s'lat, RV s' sep, TRPG, RAP, SV, CO, GLS
  Pulmonary circulation mPAP rest, mPAP low-intensity, mPAP high-intensity, mPAP/CO, mPAP/CO slope
Physical activity via Actigraph wGT3X-BT | baseline, 3 and 6 months
  PA measurement during waking hours in the period of 7 days with minimal valid time of 2 week and 2 weekend days. Total volume of PA is calculated via vector magnitude after raw data processing via GGIR script in Rstudio. Calculation of average steps/day is performed via Actilife software v6.13.5.
Body composition (%fat) via bioelectrical impedance | baseline, 3 and 6m
  Measurement of % lean and fat-mass via Bodystaat 1500 device
  Other variables:
  * waist circumference via cm tape on the level of umbilicus
  * hip circumference via cm tape on the level of major trochanter
  * body mass via analog scale
  * body height via vertical cm tape

OTHER OUTCOMES:
Questionnaires (PA and SB, diet, quality of life) | baseline and 6m
  7days questionnaire in Dutch language about the usual daily routine icnluding dietary habits, physical activity and sedentary behavior and quality of life
flow mediated dilation, blood flow and HB content | baseline and 6m
  FLow mediated dilation via flow mediated dilation device; HBO2 content via near-infrared spectroscopy on the calf;

CONTACTS AND LOCATIONS:
Locations (2):
- Belgium (2):
  - Faculty of Rehabilitation Sciences and Physiotherapy, Hasselt University, Hasselt, Belgium
  - Faculty of Movement and Rehabilitation Sciences, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No